CLINICAL TRIAL: NCT07259005
Title: Breathe Hard to Breathe Easy: Online Breathwork-Assisted Therapy for Social Anxiety
Acronym: BHBE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P154; NL87496.068.24 (Registry Identifier: Dutch Trial Register)
Record Dates: First submitted 2025-06-10; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-04

CONDITIONS: Social Anxiety
Keywords: social anxiety; breathwork; psychotherapy; breathwork-assisted psychotherapy; altered states of consciousness

STUDY DESIGN:
Intervention Model Description: The study will be conducted according to a randomized experimental between-groups design with two intervention options: HV-BAT (N=48) and SP-BAT (N=48), with the latter serving as an active control. The intervention will consist of a fully online breathwork-assisted therapy (BAT) program (HV-BAT or SP-BAT), each lasting about 3 weeks. The treatment will include two preparation session, two breathwork sessions, and two integration sessions.
  baseline (t0), before each preparation session, after each preparation session (post-p1 and post-p2), before each breathwork session, after each breathwork session (post-bw1 and post-bw2), before each integration session, after each integration session (post-int1 and post-int2), 1 week after the last integration session (t1) and 1 month after last integration session (t2).
Who Masked: Outcomes Assessor
Masking Description: A list containing one code for each prospective participant will be created. Through a randomization algorithm, a person not involved in the study will assign each code to one of the two interventions. Participants who fulfill the inclusion and do not meet the exclusion criteria will be assigned the first available code from the list. Participants will be blind to the study hypotheses and the specific technique used in the other treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathwork-assisted Therapy 1 (Experimental): The investigational treatment will include two preparation sessions, two breathwork sessions, and two integration sessions.
  Interventions: Behavioral: Breathwork-Assisted Therapy 1
- Breathwork-Assisted Therapy 2 (Active Comparator): The control treatment will include two preparation sessions, two breathwork sessions, and two integration sessions.
  Interventions: Behavioral: Breathwork-Assisted Therapy 2

INTERVENTIONS:
Behavioral: Breathwork-Assisted Therapy 1 — The investigational treatment will include two preparation sessions, two breathwork sessions, and two integration sessions.
  Arms: Breathwork-assisted Therapy 1
Behavioral: Breathwork-Assisted Therapy 2 — The comparator treatment will include two preparation sessions, two breathwork sessions, and two integration sessions.
  Arms: Breathwork-Assisted Therapy 2

SUMMARY:
This study aims to investigate the potential of supplementing psychotherapy with breathing techniques as a new online therapeutic approach to reduce social anxiety (SA). Clinically significant SA affects a substantial portion of the population (about 13%) and is associated with strong negative feelings of shame and anxiety in social settings. Such emotional distress leads to impairment in personal, relational, and professional functioning and may result in increasing degrees of social isolation.

In response to the demand for improved treatments for SA, this project aims to explore the efficacy of a novel treatment approach integrating online psychotherapy with online breathwork sessions designed to induce ASC.

We will recruit 96 individuals with SA, who will be randomly divided into two groups: one group will receive the new combined breathwork-assisted psychotherapy, and the other an active control intervention that does not induce ASC. Over the treatment duration, the effectiveness of these treatments will be closely monitored using established psychological scales and by observing patients in live interactions before and after therapy.

This project is expected to open the way to a more accessible and effective treatment option for a large group of people struggling with SA. More broadly, the findings will also contribute to our understanding of how ASC, induced through breathing techniques, can be used therapeutically. This could change the way a variety of mental health conditions (e.g., other anxiety-related conditions and depression) are treated, making a substantial impact on public health and the way mental health disorders are approached and managed.

DETAILED DESCRIPTION:
Rationale: Clinically significant social anxiety affects a substantial portion of the population (about 13%) and is associated with strong negative feelings of shame, anxiety in social settings, and significant personal, relational and professional impairment. Importantly, recent estimates suggest that between half and one-third of these individuals do not respond to conventional therapies. Recent findings show better treatment outcomes for a variety of mental health conditions when psychological treatments are complemented by sessions during which participants experience altered states of consciousness. In response to the demand for improved treatments for social anxiety, this project aims to investigate the efficacy of a novel treatment approach integrating online therapy with online breathwork sessions designed to induce altered states of consciousness.

Objective: The aim is to test online-delivered breathwork-assisted therapy to reduce social anxiety.

Study design: The study will be conducted according to a randomized, experimental, between-groups design with two breathwork-assisted therapy interventions. The intervention will consist of a total of 6 sessions including two preparation sessions, two breathwork sessions, and two integration session.

Study population: 96 adult individuals with social anxiety (Liebowitz Social Anxiety Scale score > 49).

Intervention (if applicable): Breathwork-assisted therapy 1 or breathwork-assisted therapy 2.

Main study parameters/endpoints: Primary outcomes will be self-reported levels of social anxiety. Performance and physiological response in a social interaction task will be used as a secondary measure.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participants will be invited to the lab twice for the administration of behavioral tasks and two more times to participate to the breathwork sessions. Each visit will last about 2 hours. The treatment will run online and includes activities for a total 6.5h. Finally, we estimate a cumulative 1 hour to fill in all questionnaires. The total maximum load per participant is therefore 11.5 hours. Breathwork can produce an increased state of physiological arousal accompanied by elevations in heart rate and blood pressure that are considered safe in appropriately screened individuals. It also produces altered states of consciousness that may, in some cases, be characterized by transient anxiety. Participants may also experience discomfort during the social interaction task. In case the treatment yields the expected results, a potential benefit may be the reduction of social anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in the English or Dutch language
* Aged between 18 and 65
* LSAS score ≥50
* Written informed consent

Exclusion Criteria:

* Hypotension (diastolic < 60 mmHg; systolic > 90 mmHg) or hypertension (diastolic > 90 mmHg; systolic > 140 mmHg)
* History or presence of psychotic or bipolar disorders or first-degree relatives suffering from this
* History of respiratory or cardiovascular/heart problems or disease, cerebral aneurysm
* History of fainting or syncope, epilepsy or seizures
* History of panic disorder or panic attacks,
* Having had adverse reactions with prior breathwork sessions (i.e., fainting),
* Pregnancy, thinking one might be pregnant, trying to get pregnant, or breastfeeding
* Any problems affecting the ability to pace breathing (i.e., active/chronic respiratory infection including blocked nose/cough/cold/fever, etc.), breathlessness, abnormally slow breathing (bradypnea), or abnormally fast breathing (tachypnoea), any other physical/mental health conditions or current life events impairing the ability to engage in activities involving breath control
* Taking any regular medication other than the contraceptive pill, including medications to reduce blood pressure (i.e., Ramipril or other ACE-inhibitors) and beta-blockers (i.e., Propranolol).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-04-10 (Estimated); Study Completion 2028-04-10 (Estimated)

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale | The LSAS will be administered at all study timepoints: baseline, after each treatment session, 1 week and 1 month after the end of treatment.
  The LSAS (25) is a widely recognized instrument designed to assess the severity of SA. The LSAS measures both the fear and avoidance associated with social and performance situations. It consists of 24 items, divided into two subscales: 13 items addressing social interaction situations and 11 items focusing on performance situations. Each item is rated on a Likert scale from 0 (none) to 3 (severe) for fear, and from 0 (never) to 3 (usually) for avoidance, yielding a total possible score range of 0 to 144. The scale's dual focus allows for a comprehensive assessment of SA, making it a valuable tool for both therapy settings and research.
  The LSAS has demonstrated strong psychometric properties, including high internal consistency and test-retest reliability (26). It is also sensitive to changes in symptomatology, which makes it useful for evaluating treatment outcomes (27). The scale's validity has been established through correlations with other

SECONDARY OUTCOMES:
Getting Acquainted Task | The GAT will be administered at baseline and 1 week after the last treatment session.
  The GAT is an assessment tool used to evaluate SA by observing how an individual performs in a structured social interaction (29). The participant will be paired with a confederate and asked to engage in a conversation to get to know each other. This scenario is designed to elicit behaviors and responses indicative of SA, such as difficulty initiating conversation, discomfort, or avoidance behaviors. The task will involve different confederates at the two assessment timepoints to reduce habituation effects and will be video recorded and analyzed later for social performance assessment (29, 30). The assessment will be carried out by blinded raters on two dimensions: anxious appearance (fidgeting, blushing, laughing nervously and feelings of nervousness) and social behavior (making eye contact, completing of sentences, coherence, silences, listening, showing interest, responding) (29).
Heart Rate Variability | HRV will be assessed at baseline and 1 week after the last treatment session.
  During the GAT heart-rate variability (HRV) will be assessed through the use of an ECG device.
Salivary Cortisol | SC will be assessed at baseline and 1 week after the last treatment session.
  Before, immediately after and 30 minutes after the end of the GAT, saliva samples will be collected to measure the concentration of salivary cortisol (SC).

OTHER OUTCOMES:
State and Trait Anxiety | The STAI will be administered at all study timepoints: baseline, after each treatment session, 1 week and 1 month after the end of treatment.
  State and Trait Anxiety Inventory (STAI) The State-Trait Anxiety Inventory (STAI; 66) is a widely used psychological instrument designed to measure two distinct types of anxiety: state anxiety (temporary, situational anxiety) and trait anxiety (a general tendency to experience anxiety across situations). The STAI consists of 40 self-report items, divided equally into two subscales: the State Anxiety Scale (S-Anxiety) and the Trait Anxiety Scale (T-Anxiety). Each item is rated on a 4-point Likert scale, with scores ranging from 20 to 80 for each subscale, where higher scores indicate greater levels of anxiety.
Empathy | The IRI at baseline and 1 week after the last treatment session.
  The Interpersonal Reactivity Index (IRI) (51) is a 28-item questionnaire consisting of 4 discrete seven-item scales i.e. 'Fantasy' (tendency to imaginatively transpose oneself into fictional situations), 'Perspective-Taking' (tendency to spontaneously adopt the psychological viewpoint of others), 'Empathic Concern' (taps the respondents' feelings of warmth, compassion, and concern for others), and 'Personal Distress' (assesses self-oriented feelings of anxiety and discomfort resulting from tense interpersonal settings).
Well-Being | The WHO-5 at baseline, 1 week after the last treatment session and one month after the last treatment session.
  The World Health Organisation - Well-Being Index (WHO-5) (52) is a short, self-reported measure designed to evaluate subjective well-being. The WHO-5 is widely used in therapy and research settings to assess general emotional well-being and screen for depression. The index consists of five items, each reflecting a positive aspect of mental health, such as feeling cheerful, calm, active, rested, and interested in daily life. Respondents rate each item on a 6-point Likert scale ranging from 0 (at no time) to 5 (all of the time), based on their experiences over the past two weeks.
  The total score of the WHO-5 ranges from 0 to 25, with higher scores indicating better well-being. A score below 13 suggests poor well-being. The WHO-5 is valued for its simplicity, brevity, and strong psychometric properties, including high internal consistency and sensitivity to change (52).
Resilience | The RS will be administered at baseline, 1 week after the last treatment session and one month after the last treatment session.
  The Resilience Scale (RS) is a well-validated instrument designed to measure the resilience levels of individuals, reflecting their ability to cope with stress and adversity (53). The RS aims to quantify the personal qualities that enable individuals to thrive despite challenging circumstances. The scale consists of 25 items and respondents rate each item on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree).
Cognitive flexibility | The CFI will be administered at at baseline, 1 week after the last treatment session and one month after the last treatment session.
  The Cognitive Flexibility Index (CFI) is a psychometric tool designed to measure an individual's cognitive flexibility, which refers to the mental ability to switch between thinking about different concepts and thinking about multiple concepts simultaneously (54). The CFI assesses cognitive flexibility through 20 self-report items that reflect a person's capacity to adapt to new, unexpected, or changing circumstances, and to shift their thinking and behavior accordingly.
Person Perception | The IAT will be administered at baseline, 1 week after the last treatment session and one month after the last treatment session.
  The Implicit Association Task - (IAT) is a widely used psychological assessment tool designed to measure implicit attitudes and beliefs that individuals may be unable to report (55). The IAT assesses the strength of automatic associations between mental representations of objects (concepts) and evaluations (attributes). The task involves categorizing words or images that appear on a computer screen into predefined categories as quickly as possible, which reveals underlying implicit biases based on response times.
Mood | The PANAS will be administered at baseline, before and after each treatment session, 1 week and 1 month after the end of treatment.
  The Positive and Negative Affect Schedule (PANAS) is a widely utilized self-report instrument designed to measure positive and negative affective states (63). Positive affect refers to the extent to which a person feels enthusiastic, active, and alert, whereas negative affect refers to a person's general dimension of distress and unpleasurable engagement. Respondents rate the extent to which they have experienced each particular emotion on a 5-point Likert scale ranging from 1 (very slightly or not at all) to 5 (extremely) over a specified time frame, such as the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Kim PC Kuypers, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data will be made available upon reasonable and motivated request.